CLINICAL TRIAL: NCT06464224
Title: Are the Extremes of Respiratory Efforts During Assisted Ventilation Associated With Weaning Failure in Critical Ill Patients: a Prospective Observational Study
Brief Title: Extremes of Respiratory Effort in Weaning Failure From Mechanical Ventilation: a Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, JOSE ROBERTO LAPA E SILVA, Universidade Federal do Rio de Janeiro, Universidade Federal do Rio de Janeiro
Other Study IDs: 78185823.4.0000.5249
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation Pressure High; Weaning Failure
Keywords: respiratory drive; respiratory effort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low respiratory effort: patients under low respiratory effort
  Interventions: Behavioral: low respiratory effort
- high respiratory effort: patients under high respiratory effort
  Interventions: Behavioral: high respiratory effort

INTERVENTIONS:
Behavioral: low respiratory effort — patients under respiratory effort lower than -1,5 cmH2O (P0,1) and/or -7 cmH2O (Pocc)
  Groups: low respiratory effort
Behavioral: high respiratory effort — patients under respiratory effort higher than -3,5 cmH2O (P0,1) and/or -15 cmH2O (Pocc)
  Groups: high respiratory effort

SUMMARY:
The presence of high levels of respiratory effort in patients under mechanical ventilation may worsen the adjacent lung injury even after adapting protective ventilation. Primary outcome: To evaluate the failure rate of weaning from IMV and its relationship with the lower and upper extremes of respiratory effort and the upper extreme of dynamic pulmonary stress during the first 7 days of spontaneous ventilation. Analyze the influence of these extremes based on the thresholds of Pocc, P0.1 and their derivatives Pmus, Ptp, din and MP: in relation to days off MV (in the 28-day interval); Total weaning time; Rate and time for tracheostomy; Length of stay in the ICU and hospital; In-hospital mortality rate. CAAE: 78185823.4.0000.5249. Prospective multicenter observational study, carried out in the ICUs of Glória D'or and Niteroi D'or hospitals, from January 2024 to July 2026, in patients over 18 years old, undergoing orotracheal intubation and IMV, in their first 7 days on spontaneous ventilation. Hypothesis: Extremes of respiratory effort and dynamic pulmonary stress would be associated with a higher rate of weaning from IMV, as well as longer time on IMV and subsequent longer hospital stay.

DETAILED DESCRIPTION:
Introduction: The presence of high levels of respiratory effort in patients under mechanical ventilation may worsen the adjacent lung injury even after adapting protective ventilation, potentially prolonging the MV period. Primary outcome: To evaluate the failure rate of weaning from IMV and its relationship with the lower and upper extremes of respiratory effort and the upper extreme of dynamic lung stress during the first 7 days of spontaneous ventilation. Secondary outcomes: Analyze the influence of these extremes based on the thresholds of Pocc, P0.1 and their derivatives Pmus, Ptp, din and MP: in relation to days off MV (in the 28-day interval); Total weaning time; Rate and time for tracheostomy; Length of stay in the ICU and hospital; evaluate the variation in ventilation distribution through electrical impedance tomography with the extremes of Pocc and Pmus; analyze the fraction of diaphragmatic thickening and diaphragmatic excursion through diaphragmatic ultrasound at the upper and lower levels of Pocc and Pmus; In-hospital mortality rate. Methodology: CAAE: 78185823.4.0000.5249; Prospective multicenter observational study, carried out in the ICUs of Glória D'or and Niteroi D'or Hospitals, from January 2024 to July 2026, in patients over 18 years old, undergoing orotracheal intubation and IMV, in their first 7 days on spontaneous ventilation, excluding if patients with neuromuscular disease; Phrenic nerve injury; MV for less than 24 hours; Previously tracheostomized patient; Age under 18; Use of neuromuscular blocker > 72h; COPD sufferer; Pregnancy; Patient under palliative care; COVID-19 pneumonia; Patients reintubated after extubation in this hospitalization for less than 3 weeks. Statistical analysis: the sample calculation showed an estimated value of 50 patients for two candidate predictor variables; variables will be reported as mean (SD), median (IQ 25 - 75%) or absolute and relative frequencies. The estimate of any association between variables of upper and lower extremes of effort and dynamic pulmonary stress, as well as the ventilatory parameters used will be evaluated with preliminary univariate analysis (chi-square test with Yates' correction or Fisher's exact test), followed by a model multivariate logistic regression analysis adjusted for all clinical variables at hospital admission. Survival time, as well as hospital admission time until the event, will be analyzed using Kaplan-Meier estimates; the log-rank test will be used to compare groups. Values of p < 0.05 will be considered statistically significant. Hypothesis: Extremes of respiratory effort and dynamic pulmonary stress would be associated with a higher rate of weaning from IMV, as well as longer time on IMV and subsequent longer hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, admitted to the Glória D'or hospital, undergoing orotracheal intubation and invasive mechanical ventilation, in their first 7 years on spontaneous ventilation, who accept to participate in the study by signing the free and informed consent form (or by their legal responsible).

Exclusion Criteria:

* • Neuromuscular disease;

  * Phrenic nerve injury;
  * MV for less than 24 hours;
  * Previously tracheostomized patient;
  * Age under 18;
  * Use of neuromuscular blocker > 72h;
  * COPD;
  * Patients with pulmonary fibrosis;
  * Pregnancy;
  * Patient under palliative care;
  * COVID-19 pneumonia;
  * Patients reintubated after extubation in this hospitalization for less than 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under mechanical ventilation in their first seven days in spontaneous ventilation
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
weaning rate from mechanical ventilation | 2 years
  weaning rate from mechanical ventilation (%)

SECONDARY OUTCOMES:
days outside the MV (in the 28-day interval) | 2 years
  days outside the MV (in the 28-day interval)
Total weaning time (first attempt until success) | 2 years
  Total weaning time (first attempt until success) (days)
Rate and time for tracheostomy | 2 years
  Rate and time for tracheostomy (%)
Length of stay in the ICU and hospital | 2 years
  Length of stay in the ICU and hospital (days)
In-hospital mortality rate | 2 years
  In-hospital mortality rate (%)
electrical impedance tomography | 2 years
  spontaneous breathing trial failure rate (%) evaluated by electrical impedance tomography
diaphragmatic ultrassound | 2 years
  spontaneous breathing trial failure rate (%) evaluated by diaphragmatic ultrassound

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vilaça, Study Chair — manager of Physical Therapy team; Bruno Guimarães, Study Chair — manager of physical therapy team
Locations (1):
- Gloria D'or hospital, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No